CLINICAL TRIAL: NCT00333749
Title: Phase 1 1 Study Assesing the Benefit of Pasteurized Goat Milk in Reducing Disease Severity of Young Children With Oral Ulcer Diseases
Brief Title: The Effectiveness of Pasteurized Goat Milk in the Treatment of Childhood Oral Ulcer Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dan Miron MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3870505
Record Dates: First submitted 2006-01-13; First posted 2006-06-06 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Oral Ulcer
Keywords: children
MeSH Terms: conditions — Oral Ulcer | interventions — Drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 55 children < 5 years with acute oral ulcer disease.
  Interventions: Biological: Drinking or rinsing the mouth 2-3 times for 1 day
- 2 (Placebo Comparator): 55 Children < 5 years with acute oral ulcer disease.
  Interventions: Biological: Pasturlized cow milk

INTERVENTIONS:
Biological: Drinking or rinsing the mouth 2-3 times for 1 day
  Arms: 1
Biological: Pasturlized cow milk — Drinking or rinsing the mouth 2-3 times for one day.
  Arms: 2

SUMMARY:
Children with acute diseases with oral ulcers (not included PRESENTATIONS OF SLE, IBD or IMMUNOCOMPRMIZED STATES)will receive several doses (drinking or mouth rinsing) of either pasteurized goat milk or cow milk. Children will than be followed for length of the disease - signs and symptoms.

DETAILED DESCRIPTION:
A prospective randomized controlled study that will include 110 previously health 6months - 5 years children (55 in each group) with acute oral ulcer disease (< 48 hours). Children will receive several doses (drinking or mouth rinsing) of either pasteurized goat milk or cow milk. Children will than be followed for length of the disease - sings and symptoms by questioner to parents, and physical examination by there physicians. .

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 months or < 5 years.
* Acute (< 48 hours) oral ulcer disease.
* > 5 ulcers.
* Cooperative parents .
* Signing inform consent.

Exclusion Criteria:

* All types of immunosuppression, IBD, SLE, recurrent oral ulcer, disease > 48 hours, age , 6 < months or > 5 years.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Severity of disease | 3 years
Length of disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miron, MD, Principal Investigator — HaEmek Medicak Center, Afula, Israel
Locations (1):
- Dan Miron, Afula, Israel